CLINICAL TRIAL: NCT01239537
Title: A Multi-centre, Open-label, Clinical, Phase 4 Trial, Following on From a Head-to-head Comparison Study of Two H1N1 Influenza Vaccines in Children, to Compare Firstly, the Persistence of Antibody Against the A/California/7/2009 (H1N1) Virus and Secondly the Immunogenicity and Reactogenicity of One Dose of a Non-adjuvanted Trivalent Seasonal Influenza Vaccine, in Children Who Had Received a Two-dose Immunisation Regimen of Celvapan or Pandemrix.
Brief Title: Swine Flu (Influenza A H1N1) Follow on Vaccine Study
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: 2010/03
Record Dates: First submitted 2010-11-10; First posted 2010-11-11 (Estimated); Last update posted 2017-12-08 (Actual); Status verified 2017-12

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Baxter H1N1 vaccine: Previously received 2 dose schedule of Baxter H1N1 vaccine
  Interventions: Drug: Seasonal Flu vaccine
- GSK H1N1 vaccine: Previously received 2 dose schedule of GSK H1N1 vaccine
  Interventions: Drug: Seasonal Flu vaccine

INTERVENTIONS:
Drug: Seasonal Flu vaccine — 1 dose of seasonal trivalent flu vaccine (Fluarix)

SUMMARY:
In 2009 the World Health Organization (WHO) declared the Influenza A H1N1 (swine 'flu) outbreak the first global pandemic of this century. It is thought to have been responsible for 16,226 deaths globally as of 21st February 2010. The investigators know from previous influenza outbreaks that the number of cases also tends to increase during the winter season of the years after a pandemic. There is concern that last year's pandemic influenza strain will return this winter and it has, therefore, been included in WHO's recommendations for seasonal influenza vaccine combinations.

This study will assess the duration of the immune response to the H1N1 influenza vaccines given last year, and how children will respond to this year's seasonal trivalent influenza vaccine (which includes the H1N1 strain). Participating children would receive one dose of a licensed seasonal influenza vaccine and blood tests would be taken before and after vaccination.

DETAILED DESCRIPTION:
In Autumn 2009 the investigators undertook a study assessing the safety and immunogenicity of a two-dose schedule of the two Influenza A (H1N1) vaccines purchased by the UK Government, the non-adjuvanted whole virion vaccine and the ASO3-adjuvanted split-virion, in children aged 6 months to 12 years of age. 937 children completed the study by protocol and the main findings were that the adjuvanted vaccine, while reactogenic, was more immunogenic especially in younger children (seroconversion in children under 3 years of age was 98.2% vs. 80.1%, p=0.001).

Following events in Australia, and regardless of the formal investigation outcome, it is imperative to study the reactogenicity of UK seasonal influenza vaccines in children who had previously received immunization with adjuvanted H1N1 vaccines. It would be particularly important to gain early information on the fever rates in young children in order to assess whether these are higher than expected and carry a potential risk of febrile convulsions.

It is also important to determine the immunogenicity of trivalent seasonal influenza vaccine in children previously given univalent pandemic influenza vaccine. There is emerging data that different priming strategies with adjuvanted or non-adjuvanted vaccines may lead to considerable differences in the response to subsequent influenza vaccines. In the head to head paediatric study unpublished analyses show significantly lower immunogenicity in children who had received seasonal influenza vaccines in the past, despite the receipt of two doses of either Pandemrix or Celvepan. In addition, unpublished data from a manufacturer study suggests a negative effect of two doses of Pandemrix on immune responses to subsequent seasonal vaccine when given 3 weeks after the second dose (personal communication to E Miller from MHRA). Alternatively, as shown with pandemic H5N1 influenza vaccine, there may be a significant booster response to a subsequent dose following priming 6 or 14 months previously. However, this has not been demonstrated with either Pandemrix or Celvapan, and it is unknown how previous vaccination with these vaccines will affect the immunogenicity of the H1N1 component of an unadjuvanted trivalent seasonal influenza vaccine given a year later.

The investigators therefore propose a follow-on study to compare firstly, the persistence of antibody against the A/California/7/2009 (H1N1) virus after the use of these novel H1N1 influenza vaccines and secondly the immunogenicity and reactogenicity of one dose of a non-adjuvanted trivalent seasonal influenza vaccine in children, after receiving a two-dose immunisation regimen of either Pandemrix or Celvapan.

In previous pandemics, there have been further waves of infection in the subsequent influenza seasons, particularly when the pandemic strain has drifted antigenically. It is important therefore to study the persistence of antibody against pandemic influenza A (H1N1) infection in children, particularly those for whom seasonal influenza vaccine will not be recommended next year. Should a drifted H1N1 strain emerge next season, sera from children vaccinated in 2009 with the A/California/7/2009(H1N1) strain could be used to assess the likely cross protection to such a drifted strain. The existence of this unique cohort of almost 1000 children will allow information on antibody persistence to be generated for both the non-adjuvanted whole virion vaccine (Celvapan) or the ASO3-adjuvanted split-virion vaccine (Pandemrix) and would provide a valuable source of sera to assess cross protection in the event of emergence of a drifted strain.

The investigators therefore propose a follow-on study to compare firstly, the persistence of antibody against the A/California/7/2009 (H1N1) virus after the use of these novel H1N1 influenza vaccines and secondly the immunogenicity and reactogenicity of one dose of a nonadjuvanted trivalent seasonal influenza vaccine in children, after receiving a two-dose immunisation regimen of either Pandemrix or Celvapan.

This follow-on study will also provide an important opportunity to provide data on the long term safety of the Pandemrix and Celvapan vaccines prior to enrolment in the follow-on study.

The study will use a non-adjuvanted trivalent seasonal influenza vaccine, Fluarix® (GlaxoSmithKline Biologicals, Dresden, Germany). It is approved by the EMEA for prophylaxis of influenza in all ages and has been marketed since 1987. It has consistently been shown to meet or exceed the regulatory criteria for immunogenicity against the three strains H1N1, H3N2 and B, and has a good safety profile. (18) Although the option of receiving this vaccine (and having a blood test to assess the immune response to this vaccine) will be offered to all participants in the study, participants (or parents/ guardians, on the participant's behalf) may decline to receive this vaccine and the second blood test. These participants would still be eligible to take part in the study for the first blood test assessing the persistence of antibody from the original study.

Persistence of seroprotection will be assessed by both haemagglutination inhibition (HI) and microneutralisation (MN). Although EMEA guidelines for licensure of influenza vaccine are based on HI assays, the primary objective for this study uses MN titres as its measure. The decision for the preference of MN titres over HI titres was made based on recently published observations by the Centers for Disease Control and Prevention (CDC)(19, 20) and results from the Health Protection Agency's own analysis, which showed that the MN assay generally yields higher titres and detected more seroconversions to A/California/04/2009 than the HI assay (although both generally show high correlation). The investigators therefore used MN titres as the primary outcome measure in the original NIHR funded study (Clinicaltrials.gov registration number: NCT00980850)(1)

The cellular immune response to influenza immunisation will be assessed in children where sufficient blood is available and local laboratory facilities permit. Elispot assays will be carried out using PBMCs isolated from the blood to determine the T cell response to internal influenza antigens, and haemagglutinin (pandemic H1, seasonal H1 and seasonal H3). Exploratory flow cytometry assays may also be used to determine whether the T cells are CD4+ or CD8+, and to examine cytokine secretion.

RNA expression profiles pre and post vaccination will be scrutinised in 20 participants in each group to elucidate genes that are differentially expressed in response to immunisation. This analysis could highlight genes of particular importance in vaccine responses. Furthermore, comparisons between RNA profiles and correlates of vaccine immunity may identify profiles which could be useful 'biomarkers' of vaccine induced cellular and humoral immunity in future studies.

With appropriate consent, serum samples remaining after the analyses required for this study will be stored for use in future infection and immunity related research studies at the relevant study sites.

ELIGIBILITY:
Inclusion Criteria:

The participants must have completed the original NIHR funded study (NCT00980850)(1) comparing Celvapan with Pandemrix at one of the study sites participating in this follow-on study.

A parent/legal guardian has given written informed consent after the nature of the study has been explained.

Willingness to either

1. undertake a blood test at visit 1 ('persistence' cohort)
2. complete all study procedures ('booster' cohort)

Exclusion Criteria:

Participant(s) in original study (NCT00980850)(1) who had a suspected unexpected serious adverse reaction (SUSAR).

Participants in the original study (NCT00980850)(1) who did not receive two doses of H1N1 influenza vaccine.

Participants in original study (NCT00980850)(1) who received a third dose of H1N1 influenza vaccine due to an inadequate response to two doses.

History of severe allergic reaction after previous vaccinations or hypersensitivity to any seasonal influenza vaccine component.

Current egg allergy.

Known or suspected impairment/alteration of the immune system.

Disorders of coagulation.

Immunosuppressive therapy, use of systemic corticosteroids for more than 1 week within the 3 months prior to enrolment.

Receipt of blood, blood products and/or plasma derivatives or any immunoglobulin preparation within 3 months prior to enrolment.

Previous receipt of, or intent to immunize with, any other seasonal influenza vaccine(s) throughout the 2010/2011 influenza season.

Participation in another clinical trial of an investigational medical product.

Any condition which, in the opinion of the investigator, might interfere with the evaluation of the study objectives. Children with chronic, stable medical illnesses that do not result in immunosuppression (e.g. cerebral palsy, epilepsy, cystic fibrosis, congenital heart disease) will be allowed to participate in the study, unless these conditions will in some way interfere with the completion of study procedures. Children with conditions that may alter the immune response to vaccines (e.g. Trisomy 21) or will affect the ability to accurately describe adverse events (e.g. children over 5 years of age but with severe learning difficulties) will be excluded.

Ages: 17 Months to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: We intend to recruit all interested participants who completed the original NIHR funded study (NCT00980850)(1) (n=937) into groups 1 & 2 outlined in table one above. It is anticipated that approximately 66% of these participants are likely to take part in this follow-on study; therefore the study population for groups 1 & 2 is likely to be approximately 560 children. As the option of only having a blood sample taken at visit 1 will be made available to participants in this study, there will be two cohorts of participants: the 'persistence' cohort (consenting to the baseline blood test alone) and the 'booster' cohort (consenting to the baseline blood test, seasonal influenza vaccine and post-immunisation blood test).
Sampling Method: Non-Probability Sample
Enrollment: 560 (Estimated)
Dates: Start 2010-11; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Persistence of MICRONEUTRALISING antibody titres against H1N1v | 11 - 15 months
  The percentage of children with microneutralisation (MN) titres ≥ 1:40, 11-15 months after receiving a two-dose immunisation regimen of either Celvapan or Pandemrix.

SECONDARY OUTCOMES:
Immunogenicity of trivalent seasonal influenza vaccine | 12 - 16 months
  The percentage of children who seroconvert and have a post-vaccination MN titre ≥1:40 or HI titre ≥1:32 (H1N1 strain) or who were seropositive at pre-vaccination and have a 4- fold increase in titre, following one dose of a non-adjuvanted seasonal trivalent influenza vaccine, 11-15 months after receiving a two-dose immunisation regimen of either Celvapan or Pandemrix
Reactogenicity of trivalent seasonal influenza vaccine | 12 - 16 months
  The percentage of children experiencing fever, local reactions and non-febrile systemic reactions within the 7 days following one dose of a non-adjuvanted seasonal trivalent influenza vaccine 11-15 months after receiving a two-dose immunisation regimen of either Celvapan or Pandemrix.
Persistence of antibody titres to H1N1v | 11 - 15 months
  The percentage of children with HI titre ≥ 1: 32 and the geometric mean HI and MN titres in children 11-15 months after receiving a two-dose immunisation regimen of either Celvapan or Pandemrix.
Long-term safety monitoring of Pandemrix and Celvapan | 11 - 15 months
  Specific adverse events (influenza-like illnesses (ILI), hospitalisations, febrile convulsions, autoimmunity and adverse events of special interest (AESIs) will be assessed in all participants.
T cell Responses | 11 - 15 months
  The T cell responses to internal influenza antigens and haemagglutinin (pandemic H1).
Genetics | 1 month
  The identification of genes differentially expressed in response to vaccination with the seasonal influenza strain.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Pollard, MRCP, PhD, Study Director — Oxford Vaccine Group, University of Oxford; Liz Miller, FRCPath, DSc, Principal Investigator — Public Health England; Paul Heath, FRCPCH, Principal Investigator — St George's Vaccine Institute; Adam Finn, PhD, FRCPCH, Principal Investigator — Bristol Children's Vaccine Centre; Saul Faust, MRCPCH, PhD, Principal Investigator — University of Southampton Wellcome Trust Clinical Research Facility; Matthew Snape, FRCPCH, MD, Principal Investigator — Oxford Vaccine Group; Richard Tomlinson, Principal Investigator — Royal Devon and Exeter NHS Foundation Trust
Locations (5):
- United Kingdom (5):
  - Bristol Children's Vaccine Centre, University of Bristol, Bristol
  - Royal Devon and Exeter NHS Foundation Trust, Exeter
  - St George's Vaccine Institute, University of London, London
  - Oxford Vaccine Group, University of Oxford, Oxford
  - University of Southampton Wellcome Trust Clinical Research Facility, Southampton

REFERENCES:
- [Background] de Whalley P, Walker W, Snape MD, Oeser C, Casey M, Moulsdale P, Harrill C, Andrews N, Hoschler K, Thompson B, Jones C, Chalk J, Kerridge S, Tomlinson R, Heath PT, Finn A, Faust S, Miller E, Pollard AJ. A 1-year follow-on study from a randomised, head-to-head, multicentre, open-label study of two pandemic influenza vaccines in children. Health Technol Assess. 2011 Dec;15(45):v-vi, xi-xiii, 1-128. doi: 10.3310/hta15450. PMID 22257497
- [Background] Walker WT, de Whalley P, Andrews N, Oeser C, Casey M, Michaelis L, Hoschler K, Harrill C, Moulsdale P, Thompson B, Jones C, Chalk J, Kerridge S, John TM, Okike I, Ladhani S, Tomlinson R, Heath PT, Miller E, Faust SN, Snape MD, Finn A, Pollard AJ. H1N1 antibody persistence 1 year after immunization with an adjuvanted or whole-virion pandemic vaccine and immunogenicity and reactogenicity of subsequent seasonal influenza vaccine: a multicenter follow-on study. Clin Infect Dis. 2012 Mar 1;54(5):661-9. doi: 10.1093/cid/cir905. Epub 2012 Jan 19. PMID 22267719
- [Result] Lambe T, Spencer AJ, Mullarkey CE, Antrobus RD, Yu LM, de Whalley P, Thompson BA, Jones C, Chalk J, Kerridge S, Hill AV, Snape MD, Pollard AJ, Gilbert SC. T-cell responses in children to internal influenza antigens, 1 year after immunization with pandemic H1N1 influenza vaccine, and response to revaccination with seasonal trivalent-inactivated influenza vaccine. Pediatr Infect Dis J. 2012 Jun;31(6):e86-91. doi: 10.1097/INF.0b013e318255e443. PMID 22466328